CLINICAL TRIAL: NCT01402531
Title: Submucosal Bevacizumab for the Management of Recurrent Epistaxis in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100295
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Hereditary hemorrhagic telangiectasia (HHT); nosebleed; Bevacizumab; Avastin
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Submucosal Bevacizumab (Experimental): 200mg Bevacizumab, submucosal injection
  Interventions: Drug: Submucosal Bevacizumab

INTERVENTIONS:
Drug: Submucosal Bevacizumab — 200 mg Bevacizumab, injected submucosally- 100 mg per nostril
  Other Names: Avastin

SUMMARY:
This is a research study to find out more about the use of Avastin (proper chemical name is bevacizumab) in the treatment of epistaxis (nose bleeding) in patients with Hereditary Hemorrhagic Telangiectasia (HHT).

DETAILED DESCRIPTION:
The treatment, regardless of participation in the proposed research, is to bring the patients to the operating room where under general anesthesia the nose is suctioned clean of blood clot, crust and secretion. The mucosa is then injected with a local anesthetic with adrenaline to reduce discomfort and to reduce bleeding. The nasal mucosa is treated with a KTP laser in our standard fashion. A 100mg of Avastin delivered in 4cc is then diluted with 4cc of normal saline to a total volume of 8cc. The dilution is made not for any known difference in treatment but rather it normally takes a minimum of 8cc to properly inject the nasal mucosa. The 1% Bevacizumab is then injected submucosally throughout the nasal cavity sparing the mucosa of the cartilage and the septum. The nasal cavity is then sprayed with 2cc of a fibrin sealant (EVICEL) this reduces postoperative bleeding and facilitates healing from the laser therapy. It has nothing to do with the Bevacizumab injection. The patient is then awakened and returned to the recovery room and discharged home. Beginning in approximately one week the patient is instructed to begin their hypertonic pulsatile nasal irrigations. They will follow-up in the clinic at 1 month. The data collection form is attached. Prior to treatment patient completes the HHT epistaxis severity score, blood is drawn for hematocrit, hemoglobin and serum feritin levels. Women of childbearing age all have a urine pregnancy test, required both by anesthesia and for the Bevacizumab study as well. Patients are followed monthly for the first 6 months. At 3 and 6 months the blood tests are repeated. For those living in San Diego they can be performed at UCSD. For those living outside the San Diego area they can be repeated by their primary care physician. For the ensuing 18 months patients are followed monthly either electronically or by telephone. ESS scores are calculated. Laboratory tests are not repeated. Patients are followed-up until such time as they begin re-bleeding and their ESS scores increase either above 2 or by 1 point above their 1 month post-op evaluation. Experience to date with 20 or 30 patients is that bleeding ceases within 1 to 2 weeks. Hence the 1 month score should be their optimum result. Adverse events will be recorded and appropriately reported to the IRB.

A new epistaxis severity score (ESS) has been developed and tested by the HHT Foundation. We have used this for the past several months and found it to be an excellent measure of HHT epistaxis. A copy is attached.

The minimum sample size is 10 patients. Study duration is planned for 24 months and if more patients are recruited they will be included. If fewer patients are recruited the study may be extended. Data will be reported by means and standard deviations. Patients will be compared individually and collectively to their pretreatment data specifically hematocrit, hemoglobin, serum ferritin and epistaxis severity score.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18, both male and non-pregnant females capable of making informed consent who have HHT by Curacao criteria and whose nasal bleeding due to HHT is of such a magnitude that it requires medical care.
* Females of childbearing age will be given a pregnancy test as a preliminary measure to ensure that those who become involved are not at risk.
* Generally these patients will have an ESS score of 5 or greater. However on occasion an individual with a score between 2 and 5 but not capable of cleansing their nose adequately to be involved in a Bevacizumab spray treatment may be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07-22 (Actual); Primary Completion 2013-07-27 (Actual); Study Completion 2013-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Investigator of this study passed away and we do not have the study data to upload the results.
Period: Overall Study
Arm/Group | Submucosal Bevacizumab
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Investigator of this study passed away and we do not have the study data to upload the results.
Groups:
- No Participants: The Investigator of this study passed away and we do not have the study data to upload the results.
Arm/Group | No Participants
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Epistaxis Using the Epistaxis Severity Score, Hematocrit, Hemoglobin and Serum Feritin Levels..
Description: The Investigator of this study passed away and we do not have the study data to upload the results.
Time Frame: 2 years
Population: The Investigator of this study passed away and we do not have the study data to upload the results.
Arm/Group | No Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The Investigator of this study passed away and we do not have the study data to upload the results.
Arm/Group | No Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The Investigator of this study passed away and we do not have the study data to upload the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes